CLINICAL TRIAL: NCT02382250
Title: The Relationship Between Diet, Perception of Healthy Lifestyle and the Severity of Coronary Artery Disease in Patients Referred for Coronary Angiography.
Brief Title: Relationship Between Diet, Lifestyle, and the Severity of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01623
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Dietary Habits; Coronary Artery Disease; Lifestyle
MeSH Terms: conditions — Feeding Behavior; Coronary Artery Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Catheterization Group: These are patients recruited from Bellevue Hospital and NYU Hospital Cardiac Catheterization Laboratories
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Survey will be given to all participants

SUMMARY:
This study is a prospective study of patients referred for coronary angiography at Bellevue Hospital Center and NYU Langone Medical Center. Subjects enrolled in this study will complete two one-page questionnaires, including information about diet, lifestyle, perceptions of health and perceived barriers to healthy lifestyles. Patients will be contacted at one and six months following their procedure to complete follow-up questionnaires to assess changes in diet and perceptions of their health after knowing the results of their coronary angiogram. The primary outcome measure will be change in dietary patterns/perception of lifestyle between baseline and one- month and six-month follow-up. Secondary measures will include association between dietary patterns/perception of lifestyle and degree of CAD and socioeconomic status.

DETAILED DESCRIPTION:
Purpose of the study Dietary choices are influenced by individual barriers and perceptions of health, and, therefore, information on both factors are needed to gain better insight into overall dietary health. The aim of this study is to examine if patients' knowledge of their coronary anatomy leads to dietary changes or changes in perception of health after a pre-specified follow-up time period in a ethnically, racially, and socioeconomically diverse patient population presenting for cardiac catheterization.

Study Design The proposed study is a prospective study of patients referred for coronary angiography. Subjects enrolled in this study will complete a questionnaire, including information about diet, lifestyle, perceptions of health and perceived barriers to healthy lifestyles. Demographics, information regarding medical comorbidities (including two questions on depression), baseline laboratory data (already collected for clinical purposes), and angiographic data (presence/absence of CAD and severity) will be collected. Patients will be contacted by telephone at one and six months following their procedure to complete the two one-page questionnaires again. On follow-up, patients will also be asked if they have made changes to their diet, using their completed dietary survey as a guide. Both, at baseline and on follow-up, the questionnaires will be administered verbally to be consistent. The purpose of this follow-up is to determine if a patient's knowledge of their coronary disease status affects short- and long-term changes in diet and perception of health. The primary outcome measure will be change in questionnaire response between baseline and follow-up.

Methods and Procedures Subjects for study participation will include all patients age 18 and older, referred to New York University Medical Center and Bellevue Hospital for diagnostic coronary angiography, that are able to complete the baseline questionnaire.

Consent and recruitment will be conducted in accordance of the policies of the New York University IRB and federal guidelines. For the cardiac catheterization group, the attending interventional cardiologists will be contacted to determine if a potential subject is willing to be approached for the study. Informed consent will be sought and documented from all subjects upon referral. The Principal Investigator or her appointed designee will explain the rationale, procedures and potential risks of theprocedures in the study to each participant. Each subject will be told that participation in the study described in this proposal is strictly voluntary, that refusal to participate will not alter the patient's relationship with their physician, and that the study constitutes research, that the information obtained will not be specifically helpful to the individual patient's care. After the subject has read the consent form, comprehension of the key elements of the study procedures and risks will be tested with verbal questions of the consent form content. If the subject is willing to participate, the subject will sign the IRB-approved informed consent form. Subjects will be given a copy of the consent form at the time it is obtained.

Study Technique Patients meeting the inclusion and exclusion criteria in both groups will complete two one-page questionnaires (uploaded in research navigator), one about diet and one about perceptions of health and perceived barriers to healthy lifestyles. Both of these questionnaires will be administered verbally at baseline and one- and six-month telephone follow-up. Baseline demographic information and medical information will be obtained from the patient and chart in both groups (outlined below). Information regarding medications, laboratory data, and procedural data will be obtained from the medical chart (outlined below). At the conclusion of the coronary angiography procedure, information regarding the severity of CAD will be recorded.

Data Collection

The following baseline variables will be prospectively collected:

Baseline Variables:

* Demographics including gender/race/ethnicity, body mass index, abdominal circumference, education and income level (race-ethnicity self-reported, other variables measured)
* Medical history: Previous MI, previous coronary revascularization, hypertension, diabetes mellitus, hyperlipidemia, peripheral vascular disease, previous stroke or transient ischemic attack, carotid artery or peripheral artery disease (moderate or severe or history of prior repair), and tobacco and alcohol use (collected from medical records and confirmed by patient)
* Medications: Beta blocker, diuretic, ACE-I/ARB, aspirin, thienopyridine, anticoagulants, statin, fibrates, niacin, fish oil, ezetimibe, bile acid sequestrant, glucose-lowering medications (collected from medical records and confirmed by patient)
* Laboratory data: serum creatinine, lipid panel, hemoglobin A1c, ejection fraction (normal, mild to moderately reduced, or severely reduced left ventricular systolic function) (Collected from medical records) Procedural data: (Collected from catheterization report and review of films)
* Indication for coronary angiography (determined by research team according to data provided in medical records)
* Vessels affected
* Degree of stenosis within the coronary arteries
* Post-procedural recommendations: Medical management, PCI, or coronary artery bypass surgery
* If PCI performed (collected from catheterization report):

  * Vessel treated (left main, left anterior descending, left circumflex, right coronary artery, saphenous vein graft, arterial graft) and single vessel or multivessel intervention
  * Type of lesion treated (de novo or restenotic, chronic total occlusion, long lesion, bifurcation lesion, calcification, thrombus), lesion site (ostial, proximal, mid-vessel, distal), and number of lesions treated
  * Procedural success (defined as residual stenosis <20% at the end of procedure) All electronic data will be de-identified and reside on password-protected computer. All hard copy of data will be secured in a locked cabinet in a locked office on NYU Medical Center property.

Data Analysis and Data Monitoring Results from diet and perception questionnaires will be compared between baseline and one-month and six-month follow-up using paired sample tests. This comparison will be further analyzed by degree of CAD as defined by angiographic findings. The risks associated with this study are deemed minimal. There will be no intervention or change in the care of the subjects, only data collection. Therefore, a Data Safety Monitoring Committee will not be required. The investigators will review data on a quarterly basis (or more often as necessary) to ensure the safe and proper treatment of subjects.

Subject Identification, Recruitment, and Consent Subjects will be screened and recruited when they are referred to the NYU or Bellevue cardiac catheterization laboratory for clinically indicated coronary angiography. Informed consent will be obtained by the study investigator or designated appointee prior to coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* All patients fluent in English or Spanish who are referred for coronary angiography and are fully able to fill out the baseline questionnaires.

Exclusion Criteria:

* Patients will be excluded if they 1) present with ST-segment elevation MI, 2) have previously undergone coronary revascularization, 3) do not consent or are unable to give consent, or 4) are unable to complete the baseline questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred for coronary angiography at New York University Langone Medical Center and Bellevue Hospital Center.
  Subjects will include both men and women. Every effort will be made to include equitable numbers of each gender.
  Subjects more than 18 years of age will be eligible to participate in the study. The research in question applies to the entire adult population and therefore all adults may participate.
  Subjects of any racial or ethnic background may participate in the study. There will be no enrollment restrictions based on race or ethnic origin.
  The study will not include vulnerable subjects as defined by current regulations.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Change in dietary patterns/perception of lifestyle | At time of enrollment, 1 month, 6 months

SECONDARY OUTCOMES:
Association between dietary patterns/perception of lifestyle and degree of CAD and socioeconomic status | At time of enrollment, 1 month, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, MS, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States